CLINICAL TRIAL: NCT06241781
Title: A Phase 2, Multicenter Randomized Controlled Open-label Study of Autologous Tumor Infiltrating Lymphocytes (GT101 Injection) in Patients with Recurrent or Metastatic Cervical Cancer
Brief Title: Autologous Tumor Infiltrating Lymphocytes (GT101 Injection) in Patients with Recurrent or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GT-CD-CHN-101-02
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Adult
MeSH Terms: interventions — dimethyl-2-(tetrahydro-2-furanyl)ethylsulfonium; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GT101 injection treatment group (Experimental)
  Interventions: Biological: GT101 injection
- Gemcitabine injection treatment group (Active Comparator)
  Interventions: Drug: Gemcitabine injection

INTERVENTIONS:
Biological: GT101 injection — GT101 injection to treat cervical cancer
  Arms: GT101 injection treatment group
Drug: Gemcitabine injection — Gemcitabine injection to treat cervical cancer
  Arms: Gemcitabine injection treatment group

SUMMARY:
This is a Phase II, multicenter, open-label, randomized, parallel group, treatment study to assess the efficacy and safety of Autologous Tumor Infiltrating Lymphocytes (GT101 injection) compared with Gemcitabine in participants with recurrent or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. The Patients (or legally authorized representative) Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC) ,must have the ability to understand the requirements of the study);
* 2. The patient must be 18 to 70 years of age at the time of consent;
* 3. Must have a confirmed diagnosis of malignancy of their receptive histologies or cytology: unresectable recurrent or metastatic cervical carcinomas and previously received≥ 1 prior systemic therapy;
* 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* 5. Expected survival time of ≥ 12 weeks;
* 6. Adequate normal organ and marrow function;
* 7. Before tumor resection, the confirmatory imaging of disease progress since last treatment should be documented.
* 8.Patients must have measurable disease measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria (in addition to the resected lesion).

Exclusion Criteria:

* 1.Patients with uncontrollable tumor-related pain as judged by the investigator; participants requiring painkiller must already have had a stable pain management options at the time of study entry; symptomatic lesions suitable for palliative radiotherapy should be completed prior to study entry;
* 2.Patients who have psychiatric disorders, alcohol, drug or substance abuse;
* 3.Women who are pregnant or breastfeeding, or planning to become pregnant within 1 year after cell infusion;
* 4.Participate in other clinical trials within 4 weeks prior to screening, or planning to participate in this study and other clinical trials at the same time;
* 5.Any other conditions that would make the patient unsuitable candidate for the study at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years
  Defined as time from first study treatment until disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Duration of Response | 3 years
  Defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either Progression of Disease (PD) or death due to any cause, whichever occurs first.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Safety will be monitored by incidence, nature, and severity of treatment-emergent adverse events, including adverse drug reactions graded according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - The Fifth Medical Center of the General Hospital of the People's Liberation Army of China, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Chinese Academy of Medical Sciences Cancer Hospital Shenzhen Hospital, Shenzhen, Guangdong
  - Guangxi Medical University Affiliated Cancer Hospital, Guilin, Guangxi
  - Harbin Medical University Affiliated Cancer Hospital, Ha’erbin, Heilongjjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Second Hospital of Central South University, Changsha, Hunan
  - Southeast University Affiliated Zhongda Hospital, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital Dalian University, Dalian, Liaoning
  - Dalian Medical University First Affiliated Hospital, Dalian, Liaoning
  - Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Affiliated Obstetrics and Gynecology Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan University West China Second Hospital, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yun Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No